CLINICAL TRIAL: NCT05582551
Title: Highlighting Patients At Risk for Sensory Screening (HPARSS) to Enhance Sensory Deficit Screening in Childhood Cancer Survivors
Brief Title: Patients At Risk for Sensory Screening (HPARSS) to Enhance Sensory Deficit Screening in Childhood Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202208066
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Childhood Cancer
Keywords: childhood cancer survivors; electronic medical record; sensory deficit screening; hearing loss; peripheral neuropathy; vestibular; vision
MeSH Terms: conditions — Neoplasms; Hearing Loss; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients: Highlighting Patients at Risk for Sensory Screening (HPARSS) (Experimental): * The primary oncology team will utilize the HPARSS to identify patients who are at risk for sensory deficits based on prior treatment. The HPARSS will constitute a file of that will contain eligible patients based upon their past treatment and their corresponding risk for a particular sensory deficit based upon that treatment. The patient and parent/guardian will be approached to participate in the study.
  * Sensory deficit screening will be completed in the clinic and any screening results that indicate the need for referral for diagnostic testing or therapy will be scheduled by the primary treatment team staff.
  Interventions: Other: Highlighting Patients at Risk for Sensory Screening (HPARSS)
- Providers: Highlighting Patients at Risk for Sensory Screening (HPARSS) (No Intervention): -Providers will complete a survey regarding their views of the HPARSS. The Acceptability of Intervention Measure has 4 questions and the Feasibility of Intervention Measure has 4 questions.

INTERVENTIONS:
Other: Highlighting Patients at Risk for Sensory Screening (HPARSS) — Collaborators in the Informatics Research branch of the Institute of Informatics at the Washington University School of Medicine will identify CCS at risk for sensory deficits based upon their therapy exposure to generate the HPARSS document.
  Arms: Patients: Highlighting Patients at Risk for Sensory Screening (HPARSS)

SUMMARY:
The overall goal of this study is to attempt to overcome the organizational barriers that impede prompt screening for at-risk sensory deficits in childhood cancer survivors (CCS). Using a cross sectional design study, collaborators in the Informatics Research branch of the Institute of Informatics at the Washington University School of Medicine will identify CCS at risk for sensory deficits based upon their therapy exposure to generate the highlighting patients at risk for sensory screening (HPARSS) document. The investigators will utilize the HPARSS that will link therapy related risks for sensory deficits to specific screening procedures prompting the primary oncology provider to implement screening, diagnostic testing, and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of pediatric cancer (diagnosis at <18 years of age)
* Treatment including chemotherapy and/or radiation therapy
* Completion of all cancer therapy for at least 6 months and less than 2 years
* Followed in the Division of Pediatric Hematology/Oncology Program at the Washington University School of Medicine
* Current age between 7 and 17 years of age (age where all of the screening tests are both valid and have been successfully performed by our group)
* English speaking

Exclusion Criteria:

* Undergoing active cancer treatment
* Patient under the care of the Late Effects Program at St. Louis Children's Hospital
* Received previous diagnostic testing or rehabilitative therapy for a secondary deficit eligible for screening.
* Parents and/or patient illiteracy
* No contact with treatment team in the past two years
* In foster care or without a legal guardian

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at risk for sensory deficits identified by HPARSS | Through completion of enrollment for all patients (estimated to be 9 months)
Percentage of at risk patients who fail the assigned screening test | Through completion of enrollment for all patients (estimated to be 9 months)
Percentage of patients in need of referral for screen test results who participate in formal diagnostic testing and/or treatment | Through 1 year after the completion of screening test for all participants (estimated to be 1 year and 9 months)

SECONDARY OUTCOMES:
Number and types of barriers to participation in formal diagnostic testing and therapy in CCS failing to engage in sensory screening | At approximately 2 months following the patient's screening
Number and types of facilitators to participation in formal diagnostic testing and therapy in CCS failing to engage in sensory screening | At approximately 2 months following the patient's screening
Acceptability of HPARSS as measured by the Acceptability of Intervention Measure (AIM) | To be completed at the time of enrollment completion (approximately 9 months)
  -4 questions inquiring about the acceptability of HPARSS with answers ranging from completely disagree=1 to completely agree=5. The higher the score indicates higher acceptability of the HPARSS.
Feasibility of intervention as measured by Feasibility of Intervention Measure (FIM) | To be completed at the time of enrollment completion (approximately 9 months)
  -4 questions inquiring about the feasibility of HPARSS with answers ranging from completely disagree=1 to completely agree=5. The higher the score indicates higher feasibility of the HPARSS.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hayashi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital - Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu